CLINICAL TRIAL: NCT05546996
Title: The Correlation Between FlowSense Flow Rate Measurements And: EVD Drainage Data and Intracranial Pressure (ICP) Measurements
Brief Title: EVD Drainage Data and Intracranial Pressure (ICP) Measurements
Acronym: RHAEOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Rhaeos, Inc. (Industry)
Responsible Party: Principal Investigator, Samuel McClugage, Assistant Professor- Neurosurgery, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-51840
Record Dates: First submitted 2022-08-31; First posted 2022-09-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Hydrocephalus
Keywords: EVD shunt; Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Intervention Model Description: Phase A: EVD drainage will be monitored by a digital video recorder capturing images of CSF dripping through the EVD drainage system graduated drip chamber.
  Phase B: The EVD flow rate will be measured with FlowSense over a 20-minute period (FlowSense Flow Rate) (physician and patient blinded to device data), with patients receiving standard-of-care imaging and clinical observation. Simultaneously, a digital video recorder will be used to record video of CSF dripping through the EVD drainage system graduated drip chamber.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Phase A: (No Intervention): Establish suitability of digital video recording system for quantifying CSF drainage into an EVD drainage system.
- Phase B (Other): Exploratory study to generate initial data on the correlation between FlowSense flow rate measurements (FlowSense Flow Rate) and: A) EVD drainage data, quantified via video recording; B) intracranial pressure (ICP) measurements
  Interventions: Device: FlowSense

INTERVENTIONS:
Device: FlowSense — Patients will have one or more existing external ventricular drains (EVDs). Phase B patients will additionally have an accessible (shaved) region of skin >3 cm x 3 cm overlaying the EVD tubing.
  Clinical data to be collected include: 1) total drainage volume1 over the 20-minute measurement period; 2) handheld ultrasound measurement of skin thickness2 over the EVD; and 3) an ICP waveform from a standard-of-care transducer, 4) dimensions (inner diameter and outer diameter) of tunneled catheter. Single patients may be measured multiple times during their admission; each measurement will be considered independent for analysis.
  Arms: Phase B

SUMMARY:
Rhaeos, Inc. is initially targeting hydrocephalus, a life threatening condition caused by an abnormal accumulation of cerebrospinal fluid (CSF). Implantable shunts, the gold standard treatment, often fail, leading to multiple trips to the emergency room and repeat surgeries. There is no technology available today that can easily assess CSF flow in shunts wirelessly, bedside, and without capital equipment until now.

FlowSense, is a wireless, noninvasive thermal flow sensor that can be mounted on a patient's neck overlying the shunt to detect the presence and magnitude of CSF. Similar in size to a bandage, it is composed of soft, silicone with no hard edges. Data is wirelessly transmitted to a custom designed mobile app. With FlowSense, monitoring of shunt function can occur in clinics, in-patient settings, and emergency departments, thereby reducing unnecessary imaging, hospital length of stay, and readmission costs.

DETAILED DESCRIPTION:
Hydrocephalus is caused by excess cerebrospinal fluid in the brain that can lead to lethargy, seizures, and comas. There is no cure for it nor is there any way to prevent it from happening. Affecting 1M Americans today, treatment costs the healthcare system >$2B per year. Neurosurgically implanted shunts, the standard treatment, often fail. Patients with failed shunts show nonspecific symptoms, including headaches, dizziness and nausea. CTs and MRIs are used for diagnosis, but are inconclusive, expensive, and often lead to unnecessary admissions.

Rhaeos, Inc. is a VC backed, clinical stage medical device company developing FlowSense, a patent protected platform technology and a noninvasive wireless, wearable skin patch that can assess and monitor fluid flow subdermally throughout the body. The company is initially targeting hydrocephalus, a life threatening condition caused by an abnormal accumulation of cerebrospinal fluid (CSF). Implantable shunts, the gold standard treatment, often fail, leading to multiple trips to the emergency room and repeat surgeries. There is no technology available today that can easily assess CSF flow in shunts wirelessly, bedside, and without capital equipment until now.

FlowSense, is a wireless, noninvasive thermal flow sensor that can be mounted on a patient¿s neck overlying the shunt to detect the presence and magnitude of CSF. Similar in size to a bandage, it is composed of soft, silicone with no hard edges. Data is wirelessly transmitted to a custom designed mobile app. With FlowSense, monitoring of shunt function can occur in clinics, in-patient settings, and emergency departments, thereby reducing unnecessary imaging, hospital length of stay, and readmission costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more existing external ventricular drains (EVDs).

Exclusion Criteria:

* Patients with no external ventricular drains (EVDs).

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Exploratory outcome | 1 year
  Number of participants with accurate cerebrospinal flow rate measurements (measured through the FlowSense device), EVD drainage, intracranial pressure measurements. This will be measured using a video camera. We will see the changes in flow for every 20 minutes in the recording. However, this project is not intended to be statistically powered

SECONDARY OUTCOMES:
Suitability | 1 year
  Number of times the video recording works properly by visually playing back the videos.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel McClugage, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No